CLINICAL TRIAL: NCT00759135
Title: Phase 2 Multicenter Randomized Two Dose Level and Non-Inferiority Clinical Evaluation of Transrectal Administration of NX-1207 for the Treatment of BPH
Brief Title: Phase 2 Study of NX-1207 for the Treatment of Benign Prostatic Hyperplasia (BPH) (Enlarged Prostate)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nymox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NX02-0016
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Enlarged Prostate
Keywords: Benign Prostatic Hyperplasia; BPH; Enlarged Prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — fexapotide; Finasteride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Single therapeutic dose of 2.5 mg NX-1207
  Interventions: Drug: 2.5 mg NX-1207
- 2 (Experimental): Single low dose of 0.125 mg NX-1207 for dose-response evaluation
  Interventions: Drug: 0.125 mg NX-1207
- 3 (Active Comparator): 5.0 mg finasteride q.d.
  Interventions: Drug: finasteride

INTERVENTIONS:
Drug: 2.5 mg NX-1207 — Therapeutic dose; single intraprostatic injection of 2.5 mg NX-1207
  Arms: 1
Drug: 0.125 mg NX-1207 — Low dose; single intraprostatic injection of 0.125 mg NX-1207
  Arms: 2
Drug: finasteride — Active comparator; 5.0 mg finasteride p.o. q.d. for duration of study (180 days)
  Arms: 3

SUMMARY:
This completed study evaluated the safety and efficacy of two dose levels of NX-1207 for the treatment of BPH (benign prostatic hyperplasia) versus finasteride.

DETAILED DESCRIPTION:
Subjects randomized to NX-1207 were blinded as to the dose level of NX-1207 they received.

ELIGIBILITY:
Inclusion Criteria:

1. Documented history of BPH for at least 1 year
2. AUA SI ≥ 15
3. Prostate Volume ≥ 30 mL ≤ 70 mL
4. Qmax < 15 mL/sec

Exclusion Criteria:

1. History of illness or condition that may interfere with study or endanger subject
2. Use of prescribed medications that may interfere with study or endanger subject
3. Presence of a median lobe of the prostate
4. Surgery or MIST in the previous 12 months for treatment of BPH
5. Post-void residual urine volume > 350 mL
6. PSA ≥ 10 ng/mL; prostate cancer must be ruled out for PSA ≥ 4 ng/mL

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in BPH Symptom Score (AUA SI) | 90 days

SECONDARY OUTCOMES:
Change in Prostate Volume | 90 days
Change in Qmax | 90 days
Change in BPH Symptom Score (AUA SI) | 30 days
Change in BPH Symptom Score (AUA SI) | 180 days
Number of Participants with Adverse Events, duration and severity of Adverse Events and relation, if any, to drug | 180 days

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Nymox Investigational Site, Huntsville, Alabama
  - Nymox Investigational Site, Tucson, Arizona
  - Nymox Investigational Site, Little Rock, Arkansas
  - Nymox Investigational Site, Anaheim, California
  - Nymox Investigational Site, Atherton, California
  - Nymox Investigational Site, Long Beach, California
  - Nymox Investigational Site, Modesto, California
  - Nymox Investigational Site, Newport Beach, California
  - Nymox Investigational Site, Denver, Colorado
  - Nymox Investigational Site, New Britain, Connecticut
  - Nymox Investigational Site, Sarasota, Florida
  - Nymox Investigational Site, Greenwood, Indiana
  - Nymox Investigational Site, Jeffersonville, Indiana
  - Nymox Investigational Site, Shreveport, Louisiana
  - Nymox Investigational Site, Missoula, Montana
  - Nymox Investigational Site, Las Vegas, Nevada
  - Nymox Investigational Site, Lawrenceville, New Jersey
  - Nymox Investigational Site, Marlton, New Jersey
  - Nymox Investigational Site, Voorhees Township, New Jersey
  - Nymox Investigational Site, Garden City, New York
  - Nymox Investigational Site, Poughkeepsie, New York
  - Nymox Investigational Site, Staten Island, New York
  - Nymox Investigational Site, Lancaster, Pennsylvania
  - Nymox Investigational Site, Myrtle Beach, South Carolina
  - Nymox Investigational Site, Germantown, Tennessee
  - Nymox Investigational Site, Arlington, Texas
  - Nymox Investigational Site, Brownsville, Texas
  - Nymox Investigational Site, Dallas, Texas
  - Nymox Investigational Site, McAllen, Texas
  - Nymox Investigational Site, San Antonio, Texas